| Version | Date | Changes |
|---------|----------|---------------------------------------------|
| 2.0 | 05/10/22 | 6.2; 6.3; 6.4, 6.5, 6.7, 9.1,<br>11.2, 12.1 |



# **Study Protocol**

Full Title: The return to work experiences of people with

communication disorders post-stroke: a

qualitative study

Study Acronym: ConQueSt

**Sponsor:** NHS Grampian

Sponsor Reference Number: 1-017-22

Funder: NHS Grampian Research and Development

**Endowment Research Grant** 

Chief Investigator: Emma Coutts
REC Reference Number: 22/PR/0604

**R&D Reference Number:** 2022SP001E

Version Number and Date: V2.0 5<sup>th</sup> October 2022

| The | return | to | work | experiences | of | people | with | communication | disorders | post-stroke: | а |
|---|---|---|---|---|---|---|---|---|---|---|---|
| qua | litative s | stuc | ly – Co | onQueSt | | | | | | | |

# **Signatures**

By signing this document I am confirming that I have read, understood and approve the protocol for the above study.

| Emma Coutts | | 5th October 2022 |
|--------------------|-----------|------------------|
| Chief Investigator | Signature | Date |

#### 1.0 Title

The return to work experiences of people with communication disorders post-stroke: a qualitative study

## 2.0 Summary

With an estimated incidence of 15 000 in Scotland every year, stroke is the most common cause of severe physical disability among adults in Scotland. As approximately a quarter of stroke survivors are of working age, a significant proportion of the considerable financial burden of stroke can be attributed to difficulties to returning to work because of the ensuing disabilities. Stroke-related disabilities may be obvious and physical, such as reduced mobility or limited movement in the upper limb on the affected side. However, other disabilities such as communication disorders including aphasia (language processing difficulties) and dysarthria (speech articulation difficulties) may be less apparent but equally significant, because of the importance of communication across a vast range of work activities. There has been little research into the barriers and facilitators affecting people with post-stroke communication disorders endeavoring to return to work. This study aims to address this issue by conducting semi-structured interviews with people with post-stroke communication disorders to explore their experiences of returning or attempting to return to the workplace. This study will generate important knowledge that will help inform the development of a targeted intervention for this population, which will be evaluated in a future study. It therefore represents the vital first step in understanding the problem (return to work for people with post-stroke communication disorders), which is key to the development of complex health interventions.1

## 3.0 Background and rationale

Approximately a quarter of stroke survivors are of working age,<sup>2</sup> and while estimates of return to work rates following stroke vary considerably, ranging from around 11% to 85%,3 it has been estimated that over 9 million workdays are lost in the UK alone each year because of stroke, with 26% of the total annual cost of stroke being due to loss of productivity.<sup>4</sup> In addition to the economic cost, being out of the workplace due to disability has major psychosocial costs for the individual, causing reduced social capital, sense of purpose, quality of life and standard of living. 5-6 Return to work following illness or injury is therefore an important factor in reducing these economic, social and personal consequences.7 Communication disorders resulting from a stroke are very common: an estimated 21-38% of stroke survivors are affected by aphasia (which can affect comprehension of the spoken and written word, as well as the production of speech and writing),8 and 20-30% by dysarthria.9 Because of the importance of spoken and written communication in work activities, such impairments can cause considerable barriers to return to work. 10 One review found that the return to work rate for people with post-stroke aphasia averaged 28% across the included studies, a significantly lower rate than that for the general population of working-aged stroke survivors, which was 45%.8

We recently carried out a scoping review<sup>11</sup> which found that while there has been a significant amount of research in the last ten years on factors, barriers and facilitators impacting on return to work for people following a stroke, there has been little research specific to people with post-stroke communication disorders: only two records were identified in the scoping review, one of which was a narrative review on rates of return to work<sup>8</sup> and one of which was a single case study on a person with aphasia's experiences of return to work.<sup>12</sup> Therefore, there is a need to carry out research in this area, to explore issues which are unique or particularly pertinent to people with post-stroke communication disorders. This

is especially important, given the necessity of effective communication in a wide range of work-related activities, for example as a means to engage with colleagues, to share information in order to solve problems and resolve conflicts, <sup>13</sup> and as a means to ensure health and safety. <sup>14</sup>

#### 4.0 Public involvement

People with lived experience were engaged in the design of this study and will continue to be engaged throughout its implementation. This will help to ensure that the study is relevant, the design is acceptable, the information is understandable and the results are effectively communicated at the end of the study. 15 For the design stage of the project, three people from across Scotland who were known to the Chief Investigator (CI) as having the experience of attempting to return to work with post-stroke communication disorders were contacted by letter and invited to contribute to development of this proposal. An outline of the study including the proposed research questions and methodology, written in accessible language, was sent by post or email to the two people who responded. A video call (via Microsoft Teams) was arranged with each person at least 5 days later in order for them to give their comments and make further suggestions from the perspective of their lived experience of the issue. These comments and suggestions were subsequently incorporated into the design of the study which is described below. Specific examples include explicit mention that communication refers to reading/writing as well as speech, and the inclusion of National Stroke Voices as a vehicle for recruitment. These two advisors also participated in further stages of the design, as described in the relevant sections below.

5.0 Aims and research questions

This proposed research aims to investigate the experiences of people with post-stroke

communication disorders who are attempting or have attempted to return to work. The

specific questions are:

i) What are people with post-stroke communication disorders' experiences of

attempting return to work?

ii) What barriers and facilitators are experienced by people with post-stroke

communication disorders when attempting to return to work?

iii) What do people with post-stroke communication disorders perceive their

informational and support needs to be in relation to return to work?

iv) How and by whom do people with post-stroke communication disorders perceive

that any informational and support needs could be met?

6.0 Methodology and methods

6.1 Study design

A qualitative descriptive study design will be used. This methodology seeks to discover and

understand a phenomenon from the perspectives of those experiencing it. 16 It falls within the

naturalistic approach<sup>16</sup> and attempts to interpret findings while staying close to the surface of

the data.<sup>17</sup> It is appropriate to this study because it offers the opportunity to gather rich

descriptions of a phenomenon about which little is currently known, 16 and the use of

knowledge gained may influence interventional approaches aimed at the participant

population.<sup>16</sup> Interviews will be carried out using a semi-structured format in order to allow

flexibility to explore aspects of importance to the participants while having focus maintained

by the guide guestions.18

6.2 Setting

The study will take place within Scotland. The focus will be the area covered by NHS

Grampian, NHS Greater Glasgow and Clyde, and NHS Highland health boards. Participants

can also take part from elsewhere in Scotland where they are recruited via social media or

through public adverts. This cohort is of sufficient size to make recruitment viable and

feasible, and it also represents a range of geographical areas in terms of urban/rural

classification to allow for generalizability of the findings to elsewhere in Scotland and

beyond.

6.3 Participants

Adults (aged 18 years of age and over) will be eligible for inclusion if:

they have had an ischaemic or haemorrhagic stroke (excluding Transient Ischemic

Attacks, or mini strokes) within the last 3 years

they self-identify as having communication difficulties as a result of the stroke

they were in paid employment or actively seeking work at the time of their stroke

they are attempting or have attempted (whether or not successfully) to return to paid

employment since their stroke.

Individuals will be excluded if:

they lack the capacity to consent

they are considered to have insufficient English language skills to be able to engage

effectively in an interview, given that this is a small-scale study which will not have

the resources to fund interpreter services

they have a diagnosis of a learning disability, dementia or another comorbidity
deemed to be as or more significant than the stroke in their experience of return to
work.

#### 6.4 Recruitment

Sampling will be purposive and include more than one pathway in order to recruit a wide range of participants. In one pathway, individuals will be recruited through Speech and Language Therapy services in NHS Grampian, NHS Greater Glasgow and Clyde, and NHS Highland. Speech and Language Therapists (SLTs) will identify potential participants, discuss the project with them, and give them the information pack. This pack, which was designed in consultation with the two advisors with lived experience mentioned above (Section 4.0), will include an invitation letter, Participant Information Sheet (PIS), and reply slip with a stamped addressed envelope. In a second pathway, advertising notices (again designed in consultation with the advisors mentioned in Section 4.0) will be given to groups for stroke survivors run by organisations such as the Chest Heart and Stroke Scotland and the Stroke Association across Scotland, inviting individuals to contact the research team if they wish to be considered for the study. They will then be sent an information pack including a PIS, and a reply slip with a stamped addressed envelope. In either pathway, the individual can then reply to the research team by post, email or telephone if they wish to proceed with involvement.

We will aim for a total sample size of 18 participants. We will aim to recruit 12 participants initially. If data saturation has not been reached, a further three participants will be recruited, then further groups of three until data saturation has been reached. If data saturation has been reached before 18 participants have been recruited, we will close the study early. This number is based on evidence that a sample size of 12 has been found to be the minimum for data saturation in an interview study<sup>19</sup> and also for pragmatic reasons (e.g. the predicted IRAS ID: 308674 ConQueSt/Protocol/ V2.0 5<sup>th</sup> October 2022

availability of eligible participants within the region, and the time and resource limitations of the study.) If recruitment numbers are low, a third recruitment pathway will utilise the vehicle of the National Stroke Voices public involvement group and/or social media (Twitter/Facebook accounts for relevant NHS Grampian and Robert Gordon University (RGU) departments and professional contacts of the research team). Participants will be recruited via advertisements and will be asked to contact the research team in the same way as the first and second recruitment pathways.

# 6.5 Eligibility screen and informed consent

A member of the research team will make contact with each potential participant who has consented to the initial contact or responded to an advertisement to screen against the inclusion and exclusion criteria for eligibility, discuss the study further and answer any questions about it. If the person still wishes to be involved in the study, a member of the research team will arrange to meet them at a mutually agreed venue or, where a face to face meeting is not possible, via a digital interface such as NearMe or Microsoft Teams (in the case of people recruited from the NHS Greater Glasgow and Clyde and NHS Highland areas, all meetings would be conducted via a digital interface rather than face to face). Written informed consent will be obtained before conducting the interview. The participant will initial, sign and date two copies of the consent form, one of which they will keep, the other being retained by the researcher team. Where the meeting is conducted via a digital interface,. the participant will be provided with a copy of the consent form by email or post, according to their preference, and each point will be read aloud to the participant for them to indicate their consent to participate verbally. The researcher will initial each point of the consent form as the participant agrees, and will retain this hard copy. A copy of this will be sent to the participant. This meeting would be recorded, and the recording stored (see section below on data protection).

6.6 Ineligible and non-recruited patients

Participants recruited via SLTs will have been identified as eligible by the SLTs, so it is

unlikely that they will then be found to be ineligible for inclusion when screened by a member

of the research team. It is possible however that individuals who respond to advertisements

may be found to be ineligible when screened. In this event, they will be thanked for their

interest and their time, and it will be explained to them why the current study is not

appropriate for them. They will be directed to sources of support as appropriate. A screening

log will be kept, recording how many individuals have been approached about the study;

how many individuals have contacted the research team to request an interest in

participating; and how many of these have been screened as eligible for inclusion.

As involvement will entail a single interview, it is highly unlikely that a participant would have

to be withdrawn by the research team. If a participant chooses to withdraw when data

collection has already begun (e.g. when the interview has commenced), they will be asked if

they consent to the data already collected being retained by the research team for analysis.

Their wishes in this regard will be respected.

6.7 Data collection

In the case of face to face interviews, these will be arranged with participants in a venue

suitable for them (e.g. in their own home or in a clinic or a mutually convenient community

location). The sponsor's Lone Working Policy will be adhered to, with risk assessments

carried out as appropriate, in order to reduce the risk of harm to members of the research

team. While it would be more beneficial to carry out face to face interviews because of

participants' communication problems and the potential barriers caused by digital

technology, interviews could be carried out using digital interfaces such as Microsoft Teams or NearMe if necessary. As noted above, in the case of participants recruited from NHS Greater Glasgow and Clyde and NHS Highland areas, although it would be ideal to conduct face to face interviews, this is not practical outside of the Grampian area, therefore all interviews will be conducted via a digital interface. The interview will be informed by a topic guide with items probing the overarching research questions (e.g. questions about prestroke employment/job seeking activity; feelings on considering returning to work/job seeking after stroke (especially with regard to communication problems); support from health services/third sector; discussions with employer/employment services; nature of return and adjustments made; feelings about return (especially with regard to communication problems). The topic guide questions were informed by consultation with the advisors with lived experience mentioned above (Section 4.0). In addition, they were piloted with a colleague.

The interviews will last approximately 60 minutes, but the time will vary depending on the individual and their communication needs and skills (e.g. how much information they are able to provide; whether additional time is required for them to respond to questions). Additional communication support will be given if necessary (e.g. use of writing, drawing and gesture, and communication technology). If a participant would like to take a break from the interview it can be paused, as necessary, and a further session can be arranged to complete the interview at a convenient time for the participant. Participants will be given a shopping voucher as a thank-you for taking part in the study.

The interviews will be digitally recorded on a password-protected NHS iPad (with automatic cloud storage having been disabled). The recordings will be immediately transferred onto an NHS password-protected computer and deleted from the portable device.

## 6.8 Data analysis

The audio-recordings will be transcribed by an NHS Grampian-approved transcription service. Thematic analysis will be undertaken, using the procedure outlined by Braun and Clarke. <sup>20</sup> The CI will generate the initial codes on the basis of content pertinent to the research questions. A research fellow will assist with the coding process. In order to ensure rigour, The CI, one of the collaborators (a research professor), and the research fellow will code 2-3 transcripts independently and review agreement/disagreement. This may result in refinement of the coding index and further coding and reviewing agreement, until agreement is sufficiently high for coding to be conducted by the CI or the research fellow.

An audit trail will be kept in the form of Microsoft Word documents recording discussions and decisions that are made. The data management software system NVivo will be used to facilitate data analysis. Participants will be sent a summary of the initial findings and asked if they have anything further to add. They will be able to provide this by filling in a feedback form supplied with a stamped addressed envelope. This will be an optional activity and all responses will be fully anonymous. Any additional information provided by the participants in this feedback will be incorporated into the final analysis.

# 7.0 Project management

The project will be overseen by a steering group comprised of the research team, 1-2 healthcare professionals with specialist knowledge of return to work (e.g. a vocational rehabilitation specialist and/or a physiotherapist or occupational therapist with relevant expertise) and 2-3 lay advisors with lived experience (invited from the pool of advisors who participated in the design stage, as discussed above in section 4.0). This group will meet every 3 months to discuss progress and to agree on any further decisions that require to be IRAS ID: 308674 ConQueSt/Protocol/ V2.0 5<sup>th</sup> October 2022

made during the course of the project. In keeping with current guidance, lay members will

be reimbursed for their time and travel.

A study-specific Delegation Log will be prepared, detailing the responsibilities of each

member of staff working on the study.

8.0 Inspection of records

The CI, collaborators and all institutions involved in the study shall permit study related

monitoring, audits, and Research Ethics Committee (REC) review. The CI agrees to allow

the Sponsor or, representatives of the Sponsor, direct access to all study records and source

documentation.

9.0 Good clinical practice

9.1 Ethical issues

The study will be conducted in accordance with the principles of good research practice

(GRP). In addition to Sponsorship approval, a favorable ethical opinion will be obtained from

the appropriate REC, and appropriate Research and Development (R&D) approvals will be

obtained prior to commencement of the study.

Potential participants will be given clear verbal and written information in an accessible

format (for example large font size, pictorial support) as appropriate to the nature of their

communication disorders. This information will highlight that participation is entirely voluntary

and participants can withdraw at any point without needing to give a reason and without it

affecting any healthcare or return to work support they may be receiving.

We believe that there is a low burden or risk of harm to participants. Any unexpected

distress experienced when describing the emotional impact of the stroke or any difficulties

that ensued will be minimised by sensitive and sympathetic listening, acknowledging the

distress and offering to discontinue the interview. In addition, the participant information

sheet will signpost people to sources of support, for example Chest Heart & Stroke Scotland,

or the Stroke Association.

9.2 Confidentiality

All data will be identified in a manner designed to maintain participant confidentiality. All

records will be kept in a secure storage area with limited access to study staff only. Clinical

information will not be released without the written permission of the participant, except as

necessary for monitoring and auditing by the Sponsor or its designee. The CI and study staff

involved with this study will not disclose or use for any purpose other than performance of the

study, any data, record, or other unpublished, confidential information disclosed to those

individuals for the purpose of the study. Prior written agreement from the Sponsor or its

designee will be obtained for the disclosure of any said confidential information to other

parties.

9.3 Data protection

The CI and study staff involved with this project will comply with the requirements of the

General Data Protection Regulations (GDPR) and the Data Protection Act 2018. The Health

Research Authority (HRA) recommended wording to fulfil transparency requirements under

the GDPR for health and care research has been included in the PIS.

The CI and study staff will also adhere, if appropriate, to the current version of the NHS

Scotland Code of Practice on Protecting Patient Confidentiality. Access to collated participant

data will be restricted to the CI and appropriate study staff.

Computers used to collate the data will have limited access measures via user names and

passwords.

Published results will not contain any personal data that could allow identification of individual

participants.

Participants will be assigned a code in order to de-identify them for the purposes of

transcription and analysis. A separate file containing the participants' names and contact

details will be stored separately and accessed only by the research team if necessary, e.g.

for sending the summary of initial findings or final report. All identifiable study data (i.e.

signed consent forms, the coding information with participants' details), will be stored on

password-protected NHS computers (electronic data) and/or locked filing cabinets (hard

copies consent forms) on NHS premises that are only accessible to members of the

research team and destroyed at the end of the study.

Anonymised data may be analysed on university computers as well as NHS computers

during the course of the study. This anonymised data will be transferred between institutions

using a dedicated Microsoft Teams page. Anonymised transcriptions may be printed out to

facilitate the process of data analysis. These hard copies will be stored in a locked filing

cabinet in NHS or university offices which are locked outwith working hours. Audio

recordings will be destroyed at the end of the study. Anonymised research data will be

stored for ten years in an NHS-approved storage facility.

Consent procedures will seek permission to use direct quotations from respondents. Any

identifying material (e.g. names of people/employer) will be removed from the quotation.

10.4 Insurance and indemnity

Grampian Health Board is sponsoring the study.

10.4.1 Insurance - Grampian Health Board will maintain its membership of the Clinical

Negligence and Other Risks Insurance Scheme ("CNORIS") which covers the legal liability of

Grampian in relation to the study.

**10.4.2 Indemnity:** Grampian Health Board does not provide study participants with indemnity

in relation to participation in the study but has insurance for legal liability as described above.

11.0 Output and dissemination

11.1 Authorship policy

Ownership of the data arising from this study resides with the study team and their

respective employers. Following the analysis of the study data described above in section

6.7, a final report will be prepared.

11.2 Dissemination

The findings from the study will be presented via the following channels:

Academic: a peer-reviewed manuscript in high-impact journal aimed at rehabilitation professionals and academics; a presentation at a relevant international or national

conference such as the UK Stroke Forum Conference.

**Lay**: a summary of findings provided to the study participants.

**Professional:** presentations to relevant NHS Grampian, NHS Greater Glasgow and Clyde,

and NHS Highland rehabilitation professionals involved in managing post-stroke

communication disorders and/or return to work, e.g. Occupational Therapists,

Physiotherapists, Speech and Language Therapists, Vocational Rehabilitation specialists.

As indicated above (section 2.0), the findings will be used to progress a programme of

research that will benefit people who have had a stroke. It will be combined with the findings

from our earlier scoping review11 to provide important knowledge about barriers and

facilitators to return to work for people with post-stroke communication disorders. This

knowledge will then be used in a co-production that will follow on from this study. In this co-

production, based on the facilitators identified and using strategies to overcome the barriers,

a targeted intervention will be developed to support people with post-stroke communication

disorders attempting to return to work.

12.0 Study conduct responsibilities

12.1 Protocol amendments, deviations and breaches

The CI will seek approval for any amendments to the protocol or other study documents from

the Sponsor (in the first instance), REC and NHS R&D Office(s). Amendments to the

protocol or other study documents will not be implemented without these approvals.

In the event that the CI needs to deviate from the protocol, the nature of and reasons for the

deviation will be recorded in the Clinical Report Form, documented and submitted to the

Sponsor. If this necessitates a subsequent protocol amendment, this will be submitted to the

Sponsor for approval and then to the appropriate REC and NHS R&D Office(s) for review

and approval.

In the event that a serious breach of GCP is suspected, this will be reported to the Sponsor

immediately using the form "Breach Report Form".

12.2 Study record retention

Archiving of study documents will be on NHS Grampian premises in line with the Sponsor's

Standard Operating Procedure (SOP). At the end of the study the NHS Grampian archivist will

be contacted to arrange appropriate archiving.

12.3 End of study

The end of study is defined as the last participant interview. The Sponsor, CI and/or the

steering group have the right at any time to terminate the study for clinical or administrative

reasons. The end of the study will be reported to the Sponsor and REC within 90 days, or 15

days if the study is terminated prematurely. The CI will ensure that any appropriate follow up

is arranged for all participants. A summary report of the study will be provided to the Sponsor

and REC within 1 year of the end of the study.

References

- O'Cathain A, Croot L, Duncan E, et al. Guidance on how to develop complex interventions to improve health and healthcare. BMJ Open 2019;9:e029954. doi: 10.1136/bmjopen-2019-029954
- Radford K, Grant MI, Sinclair EJ, et al. Describing return to work after stroke: a feasibility trial of 12-month outcomes. J Rehabil Med. 2020; DOI: 10.2340/16501977-2647
- Wozniak MA, Kittner SJ. Return to work after ischemic stroke: a methodological review. Neuroepidemiology. 2002;21:159–166.
- Busch MA, Coshall C, Heuschmann PU, et al. Sociodemographic differences in return to work after stroke: the South London Stroke Register (SLSR). J Neurol Neurosur PS. 2009;80:888–893.
- Clayton S, Barr B, Nylen L, et al. Effectiveness of return-to-work interventions for disabled people: a systematic review of government initiatives focused on changing the behaviour of employers. Eur J Public Health. 2012;22(3):434-439.
- Rydström I, Englund LD, Dellve L, et al. Importance of social capital at the workplace for return to work among women with a history of long-term sick leave: a cohort study. BMC Nurs. 2017;16(38) DOI 10.1186/s12912-017-0234-2
- Weerdesteijn KHN, Schaafsma F, Bonefaas-Groenewoud K, et al. Predicting return to work after long-term sickness absence with subjective health complaints: a prospective cohort study. BMC Public Health. 2020;20 DOI 10.1186/s12889-020-09203-5
- 8. Graham JR, Pereira S, Teasell R. Aphasia and return to work in younger stroke survivors. Aphasiology. 2011;25(8):952-960.
- Mitchell C, Bowen A, Tyson S, et al. Interventions for dysarthria due to stroke and other adult-acquired, non-progressive brain injury. Cochrane Database Syst Rev. 2017; (1). Available from:

- https://www.cochranelibrary.com/cdsr/doi/10.1002/14651858.CD002088.pub3/information
- 10. Niemi T, Johansson U. The lived experience of engaging in everyday occupations in persons with mild to moderate aphasia. Disabil Rehabil. 2013;35(21):1828-1834.
- 11. Coutts E, Cooper K. Interventions, barriers and facilitators associated with return to work for adults with and without communication disorders following a stroke: a scoping review. Submitted.
- 12. Morris J, Franklin S, Menger F. Returning to work with aphasia: a case study. Aphasiology. 2011;25(8):890-907.
- Bergman C, Dellve L, Skagert K. Exploring communication processes in workplace meetings: A mixed methods study in a Swedish healthcare organization. Work. 2016 Jul 26;54(3):533-541.
- 14. Alsamadani R, Hallowell M, Javernick-Will AN. Measuring and modelling safety communication in small work crews in the US using social network analysis. Construction Management and Economics. 2013;31(6):568-579.
- 15. NHS Health Research Authority. Public Involvement. Health Research Authority.

  Available from: <a href="https://www.hra.nhs.uk/planning-and-improving-research/best-practice/public-involvement/">https://www.hra.nhs.uk/planning-and-improving-research/best-practice/public-involvement/</a> [accessed 23<sup>rd</sup> September 2021].
- 16. Bradshaw, C., Atkinson, S., & Doody, O. (2017). Employing qualitative description in health care research. *Global Qualitative Nursing Research*, *4*, 1-8.
- 17. Sandelowski, M. (2000). Whatever happened to qualitative description? *Research in Nursing and Health*, 23, 334-340.
- 18. Fylan, F. (2003) Semi-structured interviewing. In J. Miles & Gilbert. P. (Eds.), A handbook of research methods for clinical and health psychology (pp. 65-78). Oxford University Press.

Guest G, Bunce A, Johnson L. How Many Interviews Are Enough?: An Experiment with Data Saturation and Variability. *Field Methods*. 2006;18(1):59-82.
 doi:10.1177/1525822X05279903

20. Braun, V., & Clarke, V. (2006). Using thematic analysis in psychology. *Qualitative Research in Psychology*, 3, 77-101.